CLINICAL TRIAL: NCT02225860
Title: Low Osmolar Diet and Adjusted Water Intake for Vasopressin Suppression in ADPKD
Brief Title: Diet as a Potential Treatment for Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11111
Record Dates: First submitted 2014-08-20; First posted 2014-08-26 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: ADPKD; Copeptin; Vasopressin; Diet; Water
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Diabetes Insipidus | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet and Water adjustment (Active Comparator): Reduction in dietary salt and protein intake
  Interventions: Behavioral: Diet and water adjustment
- Control (No Intervention): Continue with usual diet

INTERVENTIONS:
Behavioral: Diet and water adjustment — The dietary intervention consisted of three elements: low sodium (1500 mg/day), low protein (daily protein dietary allowance of 0.8 gram/kg body weight), and low urea (avoidance of preservatives, food additives, bulking agents, and chewing gum). Protein was factored by measured body weight to mirror the estimated average requirement (EAR) of healthy adults which is set on a grams per kilogram basis
  Arms: Diet and Water adjustment

SUMMARY:
The purpose of this study is to learn if dietary habits can affect vasopressin secretion in patients with autosomal dominant polycystic kidney disease. Vasopressin increases the growth of kidney cysts and accelerates disease progression. Understanding how to control secretion of this hormone based on dietary habits may help to develop treatments to control this disease. The study will include about 60 patients from Tufts Medical Center. The study will last for 2 weeks. Blood and urine tests will be done 3 times during the study period. Subjects will be randomly assigned (by chance like flipping a coin), to one of two study groups. Group 1 will be given instructions to adjust their diet. This will include adjusting the amount of water, protein, and salt intake. Group 2 will have no adjustment of diet or water. The project has tremendous public health relevance, given the large numbers of people affected by autosomal dominant polycystic kidney disease and the substantial impact of the disease on morbidity, mortality, hospitalizations,dialysis or transplant, and societal costs of caring for those patients.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common hereditary kidney disease with an estimated 600,000 persons affected in the United States and 12.5 million persons worldwide. To date, no disease-modifying treatment has been approved for the treatment of ADPKD.

Arginine vasopressin (AVP) is a key player in cyst enlargement and disease progression. It has been established that patients with ADPKD have higher levels of AVP as compared to healthy controls. Suppression, blockade or elimination of AVP slows cyst progression. AVP-V2 receptor inhibition controls disease progression in both animal models and humans, as does genetic elimination of vasopressin in the Polycystic Kidney (PCK) rat. This evidence indicates that AVP could be a promising target for therapeutic intervention. Unfortunately, the only clinically tested medication that blocks the AVP-V2 receptor (Tolvaptan) is associated with side effects including hypernatremia, hyperuricemia and elevated liver enzymes. An ideal therapeutic approach to target AVP in patients with ADPKD would be safe, easy to administer and could be adopted early in the disease process to prevent permanent kidney damage. High fluid intake presents one such possible treatment, and has been shown to suppress plasma levels of AVP, and slow cyst progression in an animal model of polycystic kidney disease. However, adherence to a high fluid intake diet is difficult to maintain in clinical practice.

To address this adherence challenge, The investigators have developed a stepwise approach of combining a low osmolar diet (low protein and salt) with adjusted water intake, with the goal of lowering the amount of water intake needed to suppress AVP secretion. The major objective of this proposal is to evaluate whether this intervention can suppress vasopressin secretion in patients with early ADPKD. Vasopressin suppression will be assessed by measuring copeptin levels, which have been shown to be a reliable surrogate marker for the circulating AVP concentration.

The rationale for this proposal is based on the fact that part of the difficulty in sustaining a low AVP level with daily water ingestion is the consumption of a diet that generates a large number of osmoles; high osmolar load stimulates vasopressin secretion to maintain water homeostasis. Hence, combining a low osmolar diet with adjusted water intake might prove to be sufficient to suppress vasopressin secretion in the clinical setting. The investigators propose the following:

Specific Aim: To conduct a randomized controlled trial to evaluate the effect of a low osmolar diet and high water intake intervention on vasopressin secretion, urine osmolality, and daily solute excretion in adult patients with ADPKD. The investigators hypothesize that a low osmolar diet combined with adjusted water intake will decrease serum copeptin level and total daily solute excretion in patients with ADPKD as compared to the control arm.

To accomplish the research goals, the current proposal builds upon existing expertise at Tufts Medical Center in conducting controlled clinical trials in patients with ADPKD.

The expected outcomes include the identification of a relevant, safe, easily tolerated and affordable intervention that can suppress vasopressin secretion in ADPKD patients early in the disease process; the proposed stepwise approach of combining a low osmolar diet and adjusted water intake carries the premise of lowering the amount of water needed to suppress AVP secretion and potentially slow the progression of this devastating disorder.

The study long-term goal is to evaluate whether this therapeutic approach could be tolerated by patients over a longer period of time, and could impact clinical outcome measures such as kidney volume and kidney function progression.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 60 years of age, who have ADPKD with an estimated glomerular filtration rate (eGFR) of 60 ml/min/1.73m2 or above

Exclusion Criteria:

1. Patients on chronic use of medications known to affect AVP secretion (Serotonin Specific Reuptake inhibitors (SSRI), Opioids, Tricyclic Antidepressants (TCA) and Tolvaptan)
2. History of diseases influencing renal concentration capacity, such as, diabetes insipidus, adrenal or thyroid deficiencies, present or prior use of lithium, or kidney diseases other than ADPKD.
3. Baseline hyponatremia (Na below 135 mEq/l)
4. Inability to comply with dietary or fluid requirements
5. Have physical or cognitive impairments which prevent participation
6. Pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Perrone, MD, Principal Investigator — Tufts Medical Center; Osama Amro, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039

RESULTS

PARTICIPANT FLOW:
Groups:
- Diet and Water Adjustment: Reduction in dietary salt and protein intake
  Diet and water adjustment
Period: Overall Study
Arm/Group | Diet and Water Adjustment | Control
Started | 17 | 17
Completed | 16 | 17
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet and Water Adjustment | Control | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Serum Copeptin From Baseline (a Reflection of Endogenous Vasopressin Production) at Week 2
Description: The copeptin level will reflect the combined effect of low osmolar diet and adjusted water intake at week 2
Time Frame: Baseline to week 2
Measure: Mean (Standard Deviation); unit: pmole/L
Arm/Group | Diet and Water Adjustment | Control
Number analyzed (Participants) | 17 | 17
pmole/L | -0.86 (1.3) | 0.39 (1.2)
Statistical Analysis 1: Comparison: Diet and Water Adjustment vs Control; The analysis of the primary and secondary outcome was based on an intention to treat principle. Copeptin was measured in each subject at baseline and week 2 and the change from baseline to end point ("delta") was calculated for all subjects. The delta copeptin between subjects in the intervention and control arms was compared with a two sample t test for independent groups. One sample t-tests of the delta were used to examine whether there was any change over time for each group separately; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

2. Secondary Outcome: Change in Total Daily Urinary Solutes From Baseline to Week 2
Description: Total daily urinary solutes (this will serve as a surrogate for diet adherence and is known to be associated with lower vasopressin secretion).
  Total daily solutes is the total amount of osmoles detected in 24 hours urine collection.
Time Frame: Baseline to week 2
Measure: Mean (Standard Deviation); unit: mOsm/Day
Arm/Group | Diet and Water Adjustment | Control
Number analyzed (Participants) | 17 | 17
mOsm/Day | -120 (212) | 27 (79)
Statistical Analysis 1: Comparison: Diet and Water Adjustment vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

3. Secondary Outcome: Change in Mean Serum Copeptin Level From Baseline to Week 1
Description: Mean serum copeptin level at week one which will reflect the effect of low osmolar diet alone.
Time Frame: baseline to week 1
Population: At week 1, there was a nonsignificant (t-test) increase in plasma copeptin to 7.1 ±5.6 in the low osmolar diet group and to 6.1 ±5.5 in the control group. The change in mean plasma copeptin level between baseline and week1 was not statistically significant between groups.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Diet and Water Adjustment | Control
Number analyzed (Participants) | 17 | 17
pmol/L | 0.9 (1.2) | 1.4 (1.3)

ADVERSE EVENTS:
Arm/Group | Diet and Water Adjustment | Control
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Small sample size and short follow up duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No